CLINICAL TRIAL: NCT00355381
Title: Evaluating Patient Information Prescriptions in Different Service Environments
Brief Title: Evaluating Patient Information Prescriptions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Library of Medicine (NLM) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JHU 04-09-03-01; 1R01LM008143 (NIH)
Record Dates: First submitted 2006-07-19; First posted 2006-07-21 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Breast Neoplasms; Premature Birth
Keywords: Information Services; Randomized Controlled Trials; Medical Records Systems, Computerized; Internet; Librarians; Breast Neoplasms; Patient Satisfaction; Health Personnel; Costs and Cost Analysis; Premature Birth
MeSH Terms: conditions — Breast Neoplasms; Premature Birth; Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Information Services (IRx) — Information services tailored to the needs of individual patients. The information prescription (IRx)or service is defined for this study as a combination of: 1)An evidence-based web site for use by patients and their families; 2) A reference interview and assistance in locating relevant general information in response to patient information needs; 3) Documentation of the questions and the information service provided in response to these in the patient's Electronic Patient Record for review by providers as needed; and, 4) Triage of patient's/parents clinical questions to providers.
  Other Names: Information prescriptions or IRx

SUMMARY:
Research shows that patient satisfaction with medical care correlates strongly with how satisfied they are with the ease of getting information from their providers regarding their medical condition. Although the Internet is a wonderful source of information for patients, research has shown that, unmediated, it comprises a potential quagmire of information poorly matched to users needs. Providers typically do not have enough time to fulfill all of their patients' information needs. One strategy to meeting the patient's information needs is to introduce librarians trained and experienced in consumer health information services into the relationship between the patient and the provider. One recently described tactic is for providers to provide information the way they of provide treatment-through an information prescription (IRx) filled by a librarian. The librarian fills the prescription by offering information services tailored to the needs of individual patients. At Johns Hopkins, we have piloted such a tactic, and in this project, extend and evaluate it. The research hypothesis is that provision of an IRx will improve patient satisfaction, provider knowledge and attitudes regarding patient information needs, and the efficiencies of care.

DETAILED DESCRIPTION:
The goal of this research is to evaluate IRx, to provide enough data so care organizations can decide whether to implement this in their own environment.

To that end, our specific aims are:

1. To evaluate the impact of IRx on patients. We are performing a randomized clinical trial, comparing IRx with standard provision of information. The primary outcome is patient satisfaction.
2. To evaluate the impact of IRx on providers. As part of the trial, provider perceptions and behavior will be assessed.
3. To evaluate the impact of IRx on the health-care system. As part of the trial, costs entailed and resources utilized will be assessed.
4. To evaluate how IRx generalizes across service environments. The trial will be performed in two environments: adult breast cancer and neonatal intensive care.

At the heart of this proposal are the randomized clinical trials. In each, patients in both intervention and control groups will receive standard clinical care in their clinic visits. Patients randomized to the intervention group will receive information services from a specially trained librarian; patients in the control groups will receive routine, current information provision. For Aim 1, immediately after their clinic visits and four weeks later, all participants will report their satisfaction on a survey that include measures of patient-provider communication. For Aim 2, participating providers are surveyed for their perceptions of information needs being met and about patient-provider interaction. For Aim 3, costs of care and costs of providing the IRx environment will be tabulated.

ELIGIBILITY:
Inclusion Criteria:

* Breast Cancer: any new patient seen in Johns Hopkins medical oncology for Breast Cancer
* Neonatal Intensive care:Biological mothers (or consenting guardians) of premature infants born and admitted or transferred in to Johns Hopkins Hospital or Bayview Medical Center neonatal intensive care units.

Exclusion Criteria:

* Breast Cancer: None
* Neonatal Intensive Care: Parents with infants whose SNAP mortality >= 80%(J Pediatr. 2001 Jan;138(1):92-100)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2004-09; Primary Completion 2008-04 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction | 4 years

SECONDARY OUTCOMES:
provider perceptions and behavior will be assessed;costs entailed and resources utilized will be assessed;how the intervention (information services) generalizes across service environments | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Nancy K Oliver, MLS, Principal Investigator — Johns Hopkins School of Medicine; Kathleen B Oliver, MLS, MPH, Study Director — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States